CLINICAL TRIAL: NCT00553423
Title: Randomized Double Blind Placebo Controlled Trial of Lactulose for the Prevention of Hepatic Encephalopathy in Cirrhotic Patients With Upper Gastrointestinal Hemorrhage
Brief Title: Lactulose for the Prevention of Hepatic Encephalopathy in Cirrhotic Patients With Upper Gastrointestinal Hemorrhage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06GS013MED
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-10

CONDITIONS: Hepatocerebral Encephalopathy; Portal-Systemic Encephalopathy; Encephalopathy, Hepatic; Encephalopathy, Hepatocerebral
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lactulose 30 ml q6h for 48 hrs
  Interventions: Drug: Lactulose
- 2 (Placebo Comparator): Placebo 30 ml q6 hrly for 48hrs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactulose — Lactulose 30 ml q6h for 48 hrs
  Arms: 1
Drug: Placebo — Placebo 30 ml q6hrly for 48 hrs
  Arms: 2

SUMMARY:
To evaluate the role of lactulose in prevention of clinically overt hepatic encephalopathy (HE) in the setting of acute upper gastrointestinal bleeding in cirrhotic patients

DETAILED DESCRIPTION:
Variceal hemorrhage occurs in 25 to 35 % of patients with cirrhosis and accounts for 80 to 90% of bleeding episodes in these patients. Around 25-30 percent of patients develop hepatic encephalopathy. Development of hepatic encephalopathy in patients with gastrointestinal bleed can cause increase morbidity with higher hospital costs in these patients. To date no randomized trial has been done in terms of prevention of encephalopathy in gastrointestinal hemorrhage. One trial has compared lactulose in combination with antibiotic against mannite, showed equal efficacy in both groups. No study has been done evaluate the efficacy of lactulose in prevention of encephalopathy in these patients.

We hypothesize that prophylactic use of Lactulose decreases the risk of development of hepatic encephalopathy with upper GI bleed in cirrhotics.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* All acute gastrointestinal bleeding in cirrhotics without hepatic encephalopathy at the time of admission in ER

Exclusion Criteria:

* Increased α-fetoprotein level/ Documented hepatoma
* Portal or hepatic vein thrombosis
* Large-volume or tense ascites requiring repeated therapeutic paracentesis
* Serious recurrent or ongoing co morbid illness (e.g., severe renal, cardiac, or respiratory failure; sepsis)
* Pregnancy
* Not willing to give consent to participate in the study
* Patients who are unable to read and write
* ER arrival time > 12 hrs from index bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2007-11; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Development of Clinically Overt Hepatic Encephalopathy | 48hours

SECONDARY OUTCOMES:
Death, hospital stay | 48hrs

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Majid, FCPS, Principal Investigator — Aga Khan University; Mohammad Salih, FCPS, Study Director — Aga Khan University; Shahid Ahmed, FCPS, Study Director — Aga Khan University; Wasim Jafri, FCPS, Study Chair — Aga Khan University
Locations (2):
- Pakistan (2):
  - Aga Khan university, Karachi, Sindh
  - Aga Khan University, Karachi, Sindh